CLINICAL TRIAL: NCT04107012
Title: Evaluation of Enamel Demineralization During Clear Aligner Orthodontic Treatment With QLF Compared to Conventional Fixed Appliances: a Randomized Clinical Trial
Brief Title: Evaluation of Enamel Demineralization During Clear Aligner Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: JUST20160295
Record Dates: First submitted 2019-07-14; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: White Spot Lesion
Keywords: White spot lesion; QLF; Clear aligners
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clear Aligner (Experimental): Group 1 treated with clear aligners
  Interventions: Device: Orthodontic treatment with clear aligner
- Fixed appliance (Active Comparator): Group 2 treated with conventional fixed appliances
  Interventions: Device: Orthodontic treatment with clear aligner

INTERVENTIONS:
Device: Orthodontic treatment with clear aligner — Included orthodontic treatment with clear aligner (eon Aligners)

SUMMARY:
Development of white spot lesions (enamel demineralization) will be evaluated quantitatively during clear aligner orthodontic treatment compared to conventional fixed appliances using quantitative light induced fluorescence (QLF)

DETAILED DESCRIPTION:
White spot lesion (WSL) may develop around fixed orthodontic appliances. With clear aligners, however, the issue is not controversial. WSL will be monitored in 2 groups of patients; one group using clear aligners and one group wearing fixed orthodontic appliances for 3 months. QLF images will be taken before treatment (T0) and 3 months after commencement of the treatment (T1). The results will be compared between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients from both genders aged (17 - 24 years).
* Class I malocclusion with mild to moderate crowding (≤ 5 mm).
* Non-extraction treatment plan.
* Optimum oral Hygiene before treatment with no signs of gingivitis and/or periodontitis.
* Maximum of 3 restored teeth.
* Absence of defective enamel formation in the form of hypocalcification or hypoplasia.

Exclusion Criteria:

-Patients with poor oral hygiene, defective enamel, extensive restorations and salivary glands diseases were excluded.

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Delta F | 3 months
  Incideance of Fluorescence loss
Lesion area | 3 months
  Incidence of the white spot lesion area

SECONDARY OUTCOMES:
Number of new lesions | 3 months
  The number of newly developed white spot lesion during orthodontic treatment
ΔR30 | 3 months
  Rate of plaque on tooth surfaces

REFERENCES:
- [Derived] Albhaisi Z, Al-Khateeb SN, Abu Alhaija ES. Enamel demineralization during clear aligner orthodontic treatment compared with fixed appliance therapy, evaluated with quantitative light-induced fluorescence: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 May;157(5):594-601. doi: 10.1016/j.ajodo.2020.01.004. PMID 32354432

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT04107012/Prot_SAP_000.pdf